CLINICAL TRIAL: NCT04439175
Title: MATCH Treatment Subprotocol I: GDC-0032 (Taselisib) in Patients With Tumors (Other Than Breast Cancer) With PIK3CA Mutation But Without KRAS Mutation or PTEN Loss
Brief Title: Testing GDC-0032 (Taselisib) as a Potential Targeted Treatment in Cancers With PIK3CA Genetic Changes (MATCH-Subprotocol I)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03142; NCI-2020-03142 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-I (Other: ECOG-ACRIN Cancer Research Group); EAY131-I (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2022-12-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (taselisib) (Experimental): Patients receive taselisib 4 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Taselisib

INTERVENTIONS:
Drug: Taselisib — Given PO
  Other Names: GDC-0032; RO5537381

SUMMARY:
This phase II MATCH treatment trial identifies the effects of GDC-0032 (taselisib) in patients whose cancer has a genetic change called PIK3CA mutation. Taselisib may stop the growth of cancer cells by blocking PIK3CA, a protein that may be needed for cell growth. Researchers hope to learn if taselisib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive taselisib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have a PIK3CA mutation as determined via the MATCH Master Protocol
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients with known left ventricular dysfunction must have echocardiogram (ECHO) or multigated acquisition scan (MUGA) within 4 weeks prior to registration to treatment and must not have left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible
* Patients must have a fasting glucose =< 125 mg/dL

  * NOTE: Please provide clear documentation that the glucose test was conducted at a fasting state
* Patients with prior treatment with an mTOR inhibitor are acceptable. These include, but are not limited to: temsirolimus, everolimus, ridaforolimus, sirolimus, CC-223, MLN128 (INK128), DS-3078, CC-115, AZD-2014, AZD8055

Exclusion Criteria:

* Patients must not have known hypersensitivity to GDC-0032 (taselisib) or compounds of similar chemical or biologic composition
* Patients must not have breast cancer
* Patients with squamous cell carcinoma of the lung who have PIK3CA mutations who have access to AND are eligible for Lung-MAP (S1400) are not eligible
* Patients must not have KRAS mutations, and/or PTEN mutation or loss, detected in the tumor sample as determined by the MATCH screening assessment. PTEN loss will be determined by immunohistochemistry
* Patients must not have had prior therapy with a PI3K inhibitor or PI3K/mTOR inhibitor. These include, but are not limited to: BEZ235, XL-765 (SAR245409), GDC-0980, PF-04691502, PF-05212384 (PKI-587), SF-1126, GSK 2126458, P-7170, BGT-226, LY3023414, GDC-0084, DS-7423, BKM-120 (buparlisib), PX-866, XL-147, GDC-0941 (pictilisib), VS-5584, BAY-80-6946, ZSTK-474, WX 037, AZD8835, GSK2636771, GS-9820, BYL719, MLN1117 (INK1117), idelalisib, TGR1202, RP6530, duvelisib (IPI-145), CUDC-907. Prior GDC-0032 (taselisib) is not allowed
* Patients must not have had prior therapy with an Akt inhibitor. These include, but are not limited to: MK-2206, GSK690693, AZD5363, triciribine, perifosine, GSK2141795, GSK2110183, SR13668, BAY1125976, GDC-0068 (ipatasertib), LY2780301, ARQ092
* Patients must not have type 1 or 2 diabetes requiring anti-hyperglycemic medication (e.g. metformin, glipizide, insulin)
* Patients must not have current dyspnea at rest or require any daily supplemental oxygen
* Patients must not have history of inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis) or active bowel inflammation (e.g. diverticulitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ian E Krop, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol I was activated on February 25, 2016. 97 patients were assigned to Subprotocol I after screening, all from the screening cohort. Of the 97 patients, 70 patients enrolled in the study between March 2016 and April 2017.
Pre-assignment Details: To be assigned to a specific MATCH subprotocol, patients needed to submit a tumor biopsy for molecular characterization and those with molecular variants addressed by treatments included in the trial entered corresponding MATCH subprotocol. For subprotocol W, patients had to have tumors with an activating PIK3CA mutation.
Groups:
- Treatment (Taselisib): Patients receive taselisib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Taselisib: Given PO
Period: Overall Study
Arm/Group | Treatment (Taselisib)
Started | 70
Started Protocol Therapy | 66
Eligible and Started Protocol Therapy (Four patients did not initiate protocol therapy and five patients initiated therapy but were subsequently found to be ineligible by central review. This is the primary analysis population.) | 61
Completed (Treatment continued until disease progression or intolerability.) | 0
Not Completed | 70
Not completed — Never started treatment | 4
Not completed — Ineligible | 5
Not completed — Adverse Event | 6
Not completed — Death | 4
Not completed — Disease progression | 44
Not completed — Withdrawal by Subject | 4
Not completed — Alternative Therapy | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Treatment (Taselisib)
Number analyzed (Participants) | 61
Age, Continuous [Median (Full Range); unit: years] | 57 [25 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 49
  More than one race | 1
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate was defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) among all eligible and treated patients. Best overall response was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. The 90% two-sided binomial exact confidence interval was calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Taselisib)
Number analyzed (Participants) | 61
percentage of participants | 0 [NA to NA] — There were no complete or partial responses.

2. Secondary Outcome: 6-Month Progression-free Survival (PFS) Rate
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. The 6-month PFS rate was estimated using the Kaplan-Meier method which can provide a point estimate for any specific time point. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS is determined
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Taselisib)
Number analyzed (Participants) | 61
percentage of participants | 19.9 [12.0 to 29.3]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Taselisib)
Number analyzed (Participants) | 61
months | 3.1 [1.8 to 3.7]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years
Description: All 70 patients enrolled to the trial were monitored for mortality, the 66 treated patients were monitored for adverse events.
Arm/Group | Treatment (Taselisib)
All-Cause Mortality (participants affected / at risk) | 66/70
Serious Adverse Events (participants affected / at risk) | 23/66
Other Adverse Events (participants affected / at risk) | 51/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Taselisib) (N=66)
Fatigue (General disorders) | 1
Sudden death NOS (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Neoplasms benign, malignant and unspecified (incl cysts and (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Taselisib) (N=66)
Anemia (Blood and lymphatic system disorders) | 8
Fatigue (General disorders) | 25
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 24
Dry mouth (Gastrointestinal disorders) | 6
Mucositis oral (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 6
Bruising (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 8
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 4
White blood cell decreased (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 18
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT04439175/Prot_001.pdf